CLINICAL TRIAL: NCT00650559
Title: Chest Wall Enlargement by Widening Sternotomy in Patients With Severe Emphysema: a Feasibility Trial.
Brief Title: Thorax Enlarging Surgery: a Novel Surgical Approach to Emphysema
Acronym: TE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: post-surgical complications in the last 2 patients
Sponsor: KU Leuven (Other)
Responsible Party: Marc Decramer, University Hospital Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TE-001; No grants or contracts
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: COPD; Emphysema
Keywords: COPD; Emphysema; thorax enlargement; LVRS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Experimental surgical intervention.
  Interventions: Procedure: Chest wall enlargement

INTERVENTIONS:
Procedure: Chest wall enlargement — Widening sternotomy
  Other Names: PEEK cages

SUMMARY:
There is a growing population of end-stage COPD patients for whom surgical treatments like lung transplantation and lung volume reduction surgery are not possible. In such patients, size mismatch between large emphysematous lungs and a restricted chest wall is a major cause for the reduction of dynamic lung volumes and consequent dyspnea. We hypothesized that enlargement of the thorax would be a potential alternative strategy to volume reduction surgery as it may improve lung mechanics by resizing the chest to the lung and does not further deprive patients from lung tissue which is already scarce.

DETAILED DESCRIPTION:
Lung volume reduction surgery primarily increases vital capacity by reducing RV more than TLC. As the chest wall is the major TLC limiting factor, an alternative approach that could circumvent size mismatch would be a surgical enlargement of the thorax cavity. Any post-operative increase of TLC would allow greater dynamic operational lung volumes to occur with an equal amount of dead space. Moreover, resizing of the thorax would have a tremendous advantage over resizing of the lung, in that it would not require resection of the lung in patients in whom lung tissue is already scarce. Chest expansion will only be guaranteed if the sternal widening osteotomy will obtain a solid union. Small poly-ether-ether-keton (PEEK) cages were designed to match both sternal halves in a 'press fit' way, which were filled with lyophilised bone and fixed with extra wires as in a classical sternotomy. These bone-filled cages function as a perfect matrix for progressive in-growth of cancellous bone.

ELIGIBILITY:
Inclusion Criteria:

patients with end-stage emphysema and

* Disabling dyspnea
* GOLD III or IV
* Residual volume > 200% predicted
* Total Lung capacity > 120% predicted
* RV/TLC > 0.6
* Resting CO2 < 50 mmHg
* diffusion capacity > 20% predicted
* age < 70 years

Exclusion Criteria:

* previous sternotomy
* contraindication of general anesthesia
* chronic treatment with corticosteroids
* any tobacco use within 6 months
* candidates for lung volume reduction surgery or lung transplantation

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2004-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Improvement of FEV1 | 1 year

SECONDARY OUTCOMES:
Improvement of exercise capacity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marc Decramer, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University hospital Leuven, Leuven, Flanders, Belgium